CLINICAL TRIAL: NCT01091844
Title: Efficacy of Retrograde Fill Vs Spontaneous FIll to Assess Voiding Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Kelly Hankins, MD - PI, Elizabeth Geller, MD - Faculty Advisor, UNC-Chapel Hill
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-1286
Record Dates: First submitted 2010-03-22; First posted 2010-03-24 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Urinary Retention; Surgery
Keywords: voiding trial, urinary retention, catheterization; Urinary retention after gynecologic surgery
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spontaneous Fill Technique (Active Comparator): We allow the bladder to spontaneously fill, then allow the patient to void and afterward catheterize the patient to check a postvoid residual ("spontaneous fill" technique").
  Interventions: Procedure: Voiding Trial
- Retrograde Fill Technique (Active Comparator): We assess bladder emptying by filling the bladder retrograde through the catheter already in place with 300 mL of saline and then removing the catheter and allowing the patient to void ("retrograde-fill" technique). We will determine postvoid residual indirectly by subtracting voided volume from the 300 mL infused volume. No catheterization will be performed with this technique unless they void less than 200 mL.
  Interventions: Procedure: Voiding Trial

INTERVENTIONS:
Procedure: Voiding Trial — After surgery, each woman will undergo a voiding trial to assess for urinary retention after surgery. This is performed on all patients undergoing surgery involving prolapse or incontinence. There are two methods commonly used to perform a voiding trial: Spontaneous Fill and Retrograde Fill techniques. Both are considered standard of care. The goal of the study is to perform both on each patient to assess their equivalency. There are no experimental interventions taking place.

SUMMARY:
Purpose: The purpose of this study is to determine if two different methods of performing a postoperative voiding trial are equivalent in evaluating urinary retention after gynecologic surgery.

Participants: The participants in this study will be women who have undergone gynecologic surgery at UNC-Chapel Hill.

DETAILED DESCRIPTION:
Subjects will be enrolled in the study when presenting to the UNC gynecology outpatient clinic for surgical preoperative evaluation. After surgery, each woman will undergo a voiding trial to assess for urinary retention after surgery. This is currently performed on all patients undergoing surgery involving prolapse or incontinence. At UNC this is usually performed by allowing the bladder to spontaneously fill, then allowing the patient to void and afterward catheterizing the patient to check a postvoid residual ("spontaneous fill" technique). In this study, we will also assess bladder emptying separately by filling the bladder retrograde through the catheter already in place with 300 mL of saline and then removing the catheter and allowing the patient to void ("retrograde-fill" technique). We will determine postvoid residual indirectly by subtracting voided volume from the 300 mL infused volume. No catheterization will be performed with this technique. Both of these techniques will be performed. The order in which the two techniques will be performed will be randomized. We will then compare the outcomes of these two techniques of voiding trials to see if they are equivalent in assessing urinary retention. Of note, the retrograde fill technique is standard at other institutions and is not considered experimental.

ELIGIBILITY:
Inclusion Criteria:

1. Women undergoing surgical correction of pelvic organ prolapse or urinary incontinence

Exclusion Criteria:

1. Unwillingness to participate in the investigation.
2. Inability to give informed consent.
3. Known preoperative voiding dysfunction
4. Plan for suprapubic catheter placement at time of surgery.
5. Age less than 18
6. Non-English speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-12; Primary Completion 2010-04 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Presence of urinary retention | Postoperative Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Hankins, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC-Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Result] Bodker B, Lose G. Postoperative urinary retention in gynecologic patients. Int Urogynecol J Pelvic Floor Dysfunct. 2003 Jun;14(2):94-7. doi: 10.1007/s00192-003-1038-3. Epub 2003 Apr 23. PMID 12851750
- [Result] Partoll LM. Efficacy of tension-free vaginal tape with other pelvic reconstructive surgery. Am J Obstet Gynecol. 2002 Jun;186(6):1292-5; discussion 1295-8. doi: 10.1067/mob.2002.123736. PMID 12066111
- [Derived] Geller EJ, Hankins KJ, Parnell BA, Robinson BL, Dunivan GC. Diagnostic accuracy of retrograde and spontaneous voiding trials for postoperative voiding dysfunction: a randomized controlled trial. Obstet Gynecol. 2011 Sep;118(3):637-642. doi: 10.1097/AOG.0b013e318229e8dd. PMID 21860294